CLINICAL TRIAL: NCT02783417
Title: Impact of Strength Training With Vascular Occlusion on the Syndrome Lipodystrophy in Patients Harboring With HIV/Aids
Brief Title: Strength Training With Vascular Occlusion in Patients Harboring With HIV/Aids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, THIAGO CÂNDIDO ALVES, Principal Investigator, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 44195315.6.0000.5393
Record Dates: First submitted 2016-05-18; First posted 2016-05-26 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Diseases
Keywords: Visceral fat
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Resistance Training with Blood Flow Restriction
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Training with vascular occlusion (Experimental): Strength Training: intensity of 30% of 1RM, with vascular occlusion pressure in members.
  Interventions: Other: Strength Training
- Traditional strength training (Experimental): Strength Training: intensity of 80% of 1RM, without vascular occlusion pressure in members
  Interventions: Other: Strength Training
- Control (No Intervention): Subject untrained.

INTERVENTIONS:
Other: Strength Training — G1: will be three series of repetitions to the concentric failure with occlusion pressure, with the two-second intervals for the concentric phase and two seconds for the eccentric phase (Moore et al., 2004;. LAURENTINO et al, 2012), with 30% of 1RM and intermittent vascular occlusion members. Will be provided one-minute intervals between sets and exercises (with the exception of the interval between the exercises of upper and lower; being provided at present a three-minute break for removal and installation of restrictive cuffs).
  G2: will be three series of repetitions to the concentric failure, with cadence of movement and intervals similar to the G1. The intensity will be 80% of 1RM without occlusion.
  Arms: Traditional strength training; Training with vascular occlusion

SUMMARY:
The use of antiretroviral therapy (ART) could prevent depression of the immune system of patients harboring with Human Immunodeficiency Virus (HIV), providing increased life expectancy, changing the classification of HIV / AIDS into a chronic illness. However prolonged use of ARTincreases the prevalence of lipodystrophy syndrome (SL), characterized by inadequate distribution of body fat and changes in lipid profile, associated with a significantly increased cardiovascular risk, among others. The practice of strength training (ST) helps in controlling SL, providing improved lipid profile and the quality of life of these patients. However, due to increased cardiovascular risk and physical weakness resulting from SL, the ST with vascular occlusion (STOV) could be a viable alternative training, to use low load (10-30% of maximal work capacity) with similar benefits ST traditional (STT), as already proven in other populations. The STOV is justified by the lower neuromuscular overhead, increasing the number of patients able to participate in this complementary therapy. The objective was to assess the impact of the combined strength training with vascular occlusion on SL and the skeletal muscle tissue in people harboring with HIV/Aids.

DETAILED DESCRIPTION:
METHODOLOGY Type of Study It is a study of the experimental type with equivalent control groups.

Sample A convenience sample will consist of approximately 60 patients seropositive for HIV / AIDS, in use of ART. Patients will be invited between routine visits in the clinic at the Special Unit for Treatment of Infectious Diseases (UETDI) of the Hospital of the Ribeirão Preto Medical School, University of São Paulo (USP HCFMRP-). They will be invited to participate voluntarily, provided that (initially) are considered eligible to participate in the study, later confirmed by medical clearance to practice physical exercises.

Place of conducting the survey:

The study will be conducted in the Orientation and Education Center of Adult and Elderly (House 5) of the Ribeirão Preto School of Nursing, University of São Paulo (EERP / USP) and UETDI HCFMRP-USP.

Lipodystrophy Syndrome (SL) The diagnosis for SL will be determined by clinical examination upon patients' reports of fat loss in the limbs, buttocks and face, with or without fat accumulation in the trunk, waist, breasts - gynecomastia (men) and cervical back, clinically confirmed by a trained professional as previously described.

Data Collection

Before the study began a medical history will be performed to determine factors that are relevant to the study and pre- and post-training, the procedures to be performed involve a number of steps involving:

* Determination Ankle Brachial Index (ABI);
* Body Composition (DC): a regional and total body analysis by examining DXA HCFMRP-USP;
* Anthropometric measurements (weight, height, skinfold thickness, perimeters and bone diameters);
* biochemical tests - to evaluate the immunological and metabolic parameters;
* Food Recall.

Index Ankle / Brachial (ITB) The ABI is calculated by the ratio of systolic blood pressure (SBP) of the posterior tibial artery or dorsalis pedis artery with higher SBP brachial or radial artery (calculated on both hemisphere). With the patient positioned supine for implementation of these measures. The PAS in both regions will be determined by means of aneroid sphygmomanometer brand "Premium®" and Doppler Vascular Portable - DV 600, brand "Martec Med®."

Body Composition The CC at the molecular levelwill be determined by scanning Total Body and Regional by DXA (Hologic®, QDR4500W software, version 11.2 QDR), being determined: bone mineral content (BMC), mass fat (MG) MG percentage (% BF) and lean soft tissue (TMM). The portion for each of these components will consider five regional sites: upper (Sup), lower (Inf), appendicular (Ape, Sup + Inf), trunk (Tro) and total (Tot). Prior to the DXA participants will be asked to empty the bladder and will wear one hospital gown. During the examination they should be positioned centrally supine on the scanner table, with outstretched legs and háluces contact; the upper body must remain extended along the trunk and hands should not be in contact with the trunk and it is important that patients stay still during the procedure.

Whereas BMC is measured by DXA bone ash of bone mass (MO) full, or approximately 95.82%, the total amount is corrected by multiplying by 1.0436 BMC. As it should be noted that although there are significant differences in the estimated BMC between DXA commercial systems, this aspect is a minimum impact on the estimate of the multicomponent CC.

Subsequently for overall changes of fat, bone and muscle tissue will be performed at processing level 2 DC components (molecular) to level 4 (organ / tissue) according to the proposed by in muscle tissue for bone tissue and into the adipose tissue, as shown in Table 1:

Table 1 - Equations of transforming the molecular level DC components to the level organ / tissue.

Magazine mass Model (kg) Skeletal Muscle TMM appendage (kg) x *1,19-1,65 Bone 1.85 x MO Adipose Tissue 1.18 x Fat Mass Body mass determined by DXA will be used for future comparisons. 3.5.3 Evaluation anthropometric Body weight and height will be determined by an electronic scale with stadiometer brand "Welmy®" featuring reading scales accurate to readings of 0.1 kg and 0.5 cm for body weight and height, respectively. Skinfolds, perimeters and bone diameters are determined by caliper, anthropometric tape and caliper with 0.1 mm reading accuracy, 0.1 cm and 0.1 mm, respectively, of the brand "Sanny Medical®".

All anthropometric measurements will be carried out according to literature recommendations.

Biochemical tests A blood sample will be collected during routine consultations for Metabolic and Immune analysis Viral Load Laboratory - Serology Sector HCFMRP-USP. The concentrations of total cholesterol (TC), triglycerides, low density lipoproteins (LDL), high density lipoprotein (HDL), insulin and fasting blood glucose are determined by an enzymatic method using the kit Wiener Lab.®. For immune responses to viral load level, when the detectable HIV RNA is> 48 cópias.mL-1. Is determined by Real Time Abbott method using the kit Siemens - Versant® HIV-1 3.0 RNA and DNA Analyzer System 340® apparatus; and CD4 + and CD8 count by flow cytometry, using Multitest® kit and Facs Calibur® cytometer (Becton Dickinson - San Jose CA).

To analyze the insulin resistance in patients, will use the homeostasis index model assessment - resistence insulin (HOMA-IR), calculated by fasting glucose formula (mmol / l = mg / dl ÷ 18) x fasting insulin (U / ml) / 22.5. The anthropometric assessment, determination of ABI and the examination of DXA will take place at HC-FMRP / USP, in a single session, at least assessors trained for each role. Laboratory tests will be performed at HC-FMRP / USP, in the morning, with all patients fasted for eight hours, the same skilled professionals during routine outpatient follow-up in UETDI HCFMRP-USP.

Protocols Strength Training (TF) Overview of Protocol

Patients will be divided into three groups, and the TF groups will be formed through the sample mirroring through the power levels:

* G1 - TFOV (n≈12; intensity of TF: 30% of 1RM). The vascular occlusion pressure members is determined individually in posterior tibial arteries and brachial or radial (computed in both hemisphere) through vascular Doppler - DV 600, the mark "Martec Med", the patient being positioned in supine and using restrictive cuffs restriction of blood flow to the brand "Missouri®" (Lower limb: 170X900 mm; Upper limb: 70X730 mm - driving cuffs).
* G2 - TFT (n≈12; TF intensity: 80% of 1RM; no vascular occlusion), and;
* G3 - Subject untrained, control group (n≈12). Individuals of G1 and G2 will undergo 12 weeks of TF, totaling 36 sessions, with weekly frequency of three times, the first two weeks of adaptation to TF.

Before each training session will be held the measurement of blood pressure (BP), heart rate (HR) and oxygen saturation in the blood (SpO2), using stethoscope and an aneroid sphygmomanometer brand "Premium®" cardiofrequency brand " Polar FT7® "and digital oximeter brand" Oximeter® ". In the absence of vital signs against indicative, begins the training protocol.

Exercises of the following: 10 minutes of heating, with the completion of five minutes on a stationary bike and a set of 15 repetitions of each exercise with heating for approximately 50% of 1RM. Thirty minutes of exercise: elbow extension in the pulley (triceps); Barbell curls (biceps); Unilateral knee flexion (hamstring) on the flexor standing; Knee extension (quadriceps) on the extensor chair, using the exercise machine station such as "Athletic 2000® Extreme" (Full Station), brand "Atletic Way®" (Porto Alegre - RS) (intensity variation 2, 5 270 kg in the independent columns); five minutes with cooling muscle relaxation.

Intensity and Volume The exercises will be distributed in two consecutive phases: Phase and Specific Adaptation Phase

Adaptation of phase (composed of six sessions for both groups):

* For groups 1 and 2, will be offered five training sessions with three sets of 12 to 15 repetitions and intensity of 50% of maximal work capacity (1RM), certain pre indirectly Adapting Stage by means of the maximum repetition test (RMs). At this stage, the concern is with respect to learning movement and speed of execution (two-second intervals for the concentric phase and two seconds for the eccentric phase). To proper adaptation of the patient to exercise.
* In the 6th training session will be given again the intensity of 1RM through the RMs test (Brzycki, 1993), to see change in the maximum force during the adaptation phase and determining the training intensity for Specific Phase. This procedure will be repeated at the 15th session of the specific period to adjust the intensity and the 30th session to verify the change of the maximum force at the end of the intervention period.

Specific phase (consisting of 30 sessions for both groups):

* G1: the first week (three sessions) will be three sets of 10 repetitions for adaptation occlusion pressure, and in the other three sessions of repetitions until concentric failure, with the two-second intervals for the concentric phase and two seconds for the eccentric phase, with 30% of 1RM and intermittent vascular occlusion members (occlusion used only during the course of the series, being released blood flow during breaks ). Will be provided one-minute intervals between sets and exercises (with the exception of the interval between the exercises of upper and lower; being provided at present a three-minute break for removal and installation of restrictive cuffs).
* G2: will be three series of repetitions to the concentric failure, with cadence of movement and intervals similar to the G1. The intensity will be 80% of 1RM without occlusion.
* The G3 not attend the TF, but will be considered as a control group, taking part only of the pre and post intervention assessments.

In order to increase security for both types of training, HR and BP patients will be monitored throughout the training session period (between exercises and series). The FC will be monitored by a heart rate monitor brand "Polar FT7® placed before the training session and the PA by a stethoscope and an aneroid sphygmomanometer brand" Premium® "that will be placed at the end of each series. As the PA will be given between 20 and 30 seconds after completion of the last rep. Before any physiological disorder or complaint, the training will be stopped and the necessary precautions and measures will be taken.

Statistical Analysis An exploratory analysis will be used to check the behavior of the data by normality test (Shapiro-Wilks) to indicate the statistical analysis of the study variables. The values (central tendency) descriptive of the morphological, metabolic and immunological characteristics will be presented in the periods (pre- and post-intervention), variance between groups and their significance levels. ANOVA (or Friedman test) to two factors will be used for comparisons between groups and moments (pre and post) concerned. All analyzes will be performed using the SPSS 17.0 software, assuming prior statistical significance of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

After agreeing to participate in the study, patients will be interviewed and so they can be included, must meet the following criteria:

* be seropositive for HIV / AIDS and not pregnant;
* Present picture of SL;
* Aged 30-60 years (both male and female);
* Using ART, with unchanged medication in the last six months;
* With stable body weight (less than 10% change in the last six months) (DOS SANTOS, WLALDEMIR ROBERTO et al, 2013.);
* Do not present Peripheral Arterial Disease, determined by the ankle / brachial index (ABI) of less than 0.91 or greater than 1.30 (Giollo Junior, 2010);
* Who are not engaged in systematic programs of physical exercise for at least three months;
* What express voluntary agreement by signing the Informed Consent and Informed (IC).

Exclusion Criteria:

They will be excluded from the study patients who:

* have any symptoms that indicate to their stay in the training program, or arising risks by doing exercises;
* miss more than six (06) training sessions not consecutively (> 15% of the sessions) (Smart et al 2014.);
* Present framework hypertensive (blood pressure greater than 140/90 mmHg from home) during the program (Noble, 2010; NHS, 2011; MANINI et al, 2012.);
* Pass the present high risk factors for thromboembolism (MOTYKIE et al., 2000; CAPRINI, 2005); CD4 + lower levels than 200 cells / mm3 (SAIF; BONA; GREENBERG, 2001; Klein et al., 2005; CRUM-Cianflone; Weekes; BAVARO, 2008; SILVA; MORI; Guimarães, 2012), and high viral load, greater than 100,000 RNA copies / mL (CRUM-Cianflone; Weekes; BAVARO, 2008; SILVA; MORI; Guimarães, 2012); concurrent diseases classified as (1) infection (Mycobacterium avium, cytomegalovirus, Pneumocystis carinii pneumonia, the herpes simplex virus, Tuberculosis, Toxoplasmosis); (2) neoplasms (Kaposi's sarcoma, non-Hodgkin's lymphoma, Hodgkin's lymphoma), (3) autoimmune diseases (Hemolytic Anemia Autoimmune - (SAIF; BONA; GREENBERG, 2001); and (5) Ischemic Heart Disease, Aortic Stenosis Severe Obstructive Hypertrophic Cardiomyopathy and (Nakajima et al., 2006).

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-08; Primary Completion 2017-02 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
strength | "pre" and "after" to "Baseline and 12 weeks"
  weight lifted in kg

SECONDARY OUTCOMES:
Body composition | "pre" and "after" to "Baseline and 12 weeks"
  kilogram (kg)

CONTACTS AND LOCATIONS:
Locations (1):
- USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alves TC, Pugliesi Abdalla P, Bohn L, Da Silva LSL, Dos Santos AP, Tasinafo Junior MF, Rossini Venturini AC, Mota J, Lopes Machado DR. Acute and chronic cardiometabolic responses induced by resistance training with blood flow restriction in HIV patients. Sci Rep. 2022 Oct 10;12(1):16989. doi: 10.1038/s41598-022-19857-3. PMID 36216952
- [Derived] Alves TC, Santos AP, Abdalla PP, Venturini ACR, Angelotti PS, Borges FG, Reis HDO, Bollela VR, Mota J, Machado DRL. Resistance training with blood flow restriction: Impact on the muscle strength and body composition in people living with HIV/AIDS. Eur J Sport Sci. 2021 Mar;21(3):450-459. doi: 10.1080/17461391.2020.1757765. Epub 2020 May 14. PMID 32349629